CLINICAL TRIAL: NCT02750007
Title: Open-label, Non-randomized, Weekly-dose Titration Study to Assess the Tolerability to HS-20004 in Type 2 (Diabetes Mellitus) Diabetic Patients
Brief Title: Tolerability to HS-20004 With Titration Administration in Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20004-Id
Record Dates: First submitted 2016-04-11; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Weekly-dose titration from 0.04mg/day HS-20004 to the maximum tolerable dose or of the ultimate 0.18mg/day
  Interventions: Drug: HS-20004

INTERVENTIONS:
Drug: HS-20004

SUMMARY:
This study is conducted in China. The aim of this trial is to assess the tolerability to HS-20004 with titration administration in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed for more than 3 months;
* HbA1c between ≥6.0 and ≤9.0 %, and FPG between ≥7.0 and ≤13.9 mmol/L;
* Body Mass Index (BMI) between 18.5 and 30 kg/m^2 (inclusive) with a total body weight of at least 50 kg;
* Agree to stop any other drugs for diabetes during washout and study period;

Exclusion Criteria:

* Treatment of GLP-1 analogues, DPP-IV enzyme inhibitors or other analogues before;
* History or family history of drug allergy;
* Smoker or alcohol abuse;
* Currently use or plan to use systemic corticosteroid;
* History of recurrent severe hypoglycemia;
* History of proliferative retinopathy or maculopathy which required acute treatment;
* Impaired hepatic or renal function, or cardiac problem;
* Uncontrolled active or untreated hypertension;
* Family history of thyroid cancer or submandibular gland cancer, or past history of pancreatitis, cholelithiasis, or serious unconscious hypoglycemia history;
* Positive of hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody;
* Subject has participated in any investigational study within 3 months, or is currently participating in another clinical study;
* Female subject of childbearing potential who does not use an acceptable method of birth control, is pregnant or planning a pregnancy, or breastfeeding, or male subject who does not use an acceptable method of birth control, within six months before randomization; Subject who cannot refrain from smoking, eating and/or drinking containing xanthine/caffeine, or strenuous exercise, or others that affect drug absorption, distribution, metabolism and excretion within 2 days before the study drug administration;
* Have any other medical abnormality (such as cardiovascular, hepatic, renal, gastrointestinal, immunologic, hematological, hormonal, metabolic, neoplasmatic or mental disease), which in the opinion of the investigator, might affect the absorption, distribution, metabolism, and excretion of the study drug, or prevent the patient from following and completing the protocol；
* Subject was not used for the study as determined by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events(TEAEs) | through study completion, an maximum of 8 weeks

SECONDARY OUTCOMES:
Number of Nausea and vomiting during titration | through study completion, an maximum of 8 weeks
Mean Change From Baseline in Body Weight at different dose steps | through study completion, an maximum of 8 weeks
Change in plasma concentration of HS-20004 from baseline at different dose steps | through study completion, an maximum of 8 weeks
Change in plasma concentration of glucose from baseline at different dose steps | through study completion, an maximum of 8 weeks
Change in plasma concentration of insulin from baseline at different dose steps | through study completion, an maximum of 8 weeks
Change in plasma concentration of glucagon from baseline at different dose steps | through study completion, an maximum of 8 weeks
The minimum dose of HS-20004 that could keep plasma glucose under 6.1 mmol/L in Type 2 Diabetic Patients | through study completion, an maximum of 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No